CLINICAL TRIAL: NCT05307627
Title: The Effects of Low Dose Naltrexone (LDN) on Diseases of Aging - A Retrospective Cross-sectional Study Into Off-label Use of LDN
Brief Title: The Effects of Low Dose Naltrexone (LDN) on Diseases of Aging
Status: Withdrawn | Type: Observational
Why Stopped: Technological barriers are affecting the participant response experience.
Sponsor: AgelessRx (Industry)
Responsible Party: Sponsor
Other Study IDs: ALRx002
Record Dates: First submitted 2022-03-07; First posted 2022-04-01 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Aging
Keywords: low-dose naltrexone; longevity; health status; quality of life
MeSH Terms: interventions — Naltrexone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Long-term (>5 years) LDN users: Participants who have been using LDN for over 5 years
  Interventions: Drug: low-dose naltrexone
- intermediate-term (1-5 years) LDN users: Participants who have been using LDN for at least 1 year, but shorter than 5 years.
  Interventions: Drug: low-dose naltrexone
- short-term (<12 months) LDN users: Participants who have been using LDN for less than a year. This group will serve as the control group.
  Interventions: Drug: low-dose naltrexone

INTERVENTIONS:
Drug: low-dose naltrexone — LDN doses <20 mg/day
  Other Names: LDN

SUMMARY:
This retrospective, observational study will assess the health status of short- and long-term low-dose naltrexone (LDN) users.

DETAILED DESCRIPTION:
Long-term (>5 years), intermediate-term (1-5 years), and short-term low-dose naltrexone (LDN) users (<12 months) will be contacted for a retrospective, observational assessment of their health status. Participants will be asked to complete a series of questionnaires assessing their quality of life, general physical and mental health, family history, the occurrence of age-related diseases, and immune status. Additionally, blood tests for immune and longevity markers will be optional for a subset of participants.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 18-120)
* Any sex
* Any ethnicity
* Taking LDN
* Willing to complete health questionnaires
* Technologically competent to complete web forms
* Subgroup: willing to undergo blood testing

Exclusion Criteria:

* LDN doses over 20 mg/day
* Terminal cancer patients (defined as stage IV and/or with a life expectancy of 12 months or less)

Ages: 18 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible long-term (>5 years), intermediate-term (1-5 years), and short-term (<12 months) LDN users
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Quality of life score | At enrollment
  The short-form (SF)-36 Questionnaire generates scores in the categories: physical function, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health. Scores up to maximum 100, with higher scores representing better quality of life
Immune Status | At enrollment
  Immune Status Questionnaire (ISQ) to define a measure of perceived immune status, consists of seven representative immune-associated symptoms and diseases. The Immune Status Questionnaire scores respondents out of 10, with 10 being a better outcome and lower scores worse outcome.

SECONDARY OUTCOMES:
General health and family history | At enrollment
  Standard questions assessing family history, and information about the dosing, duration of use, reasons for taking LDN, age, sex, weight, length, smoking and alcohol use history, substance abuse history, physical activity, other medications, and side effects of the drug, and other questions related to health and medical history.
Levine's phenotypic age | At enrollment
  Levine's phenotypic age will be calculated on basis of blood markers for age-associated diseases (glucoregulatory markers, lipids), as well as markers of inflammation
CD4/CD8 ratio | At enrollment
  Peripheral blood CD4 vs CD8 T cell ratio in cells/mm3
CMV IgG | At enrollment
  Peripheral blood cytomegalovirus (CMV) IgG antibodies in U/mL
hsCRP | At enrollment
  Peripheral blood human serum C-reactive protein (hsCRP) concentration in mg/L
IL-6 | At enrollment
  Peripheral blood serum interleukin-6 (IL-6) concentration in pg/L
TNFɑ | At enrollment
  Peripheral blood serum tumor-necrosis factor alpha (TNFɑ) concentration in pg/L
Methylation age clock testing | At enrollment
  DNA methylation array of a blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Sajad Zalzala, MD, Principal Investigator — AgelessRx
Locations (1):
- AgelessRx, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided